CLINICAL TRIAL: NCT01957475
Title: Investigation of Two Newly Developed 2-piece Convex Baseplates in Subjects With Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CP240
Record Dates: First submitted 2013-08-06; First posted 2013-10-08 (Estimated); Results first posted 2014-08-11 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Stoma - Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Coloplast Test product Z; then Coloplast Test product Y (Experimental): The subjects first test Coloplast Test product Z and after cross-over Coloplast Test product Y
  Interventions: Device: Coloplast Test product Y; Device: Coloplast Test product Z
- First Coloplast Test product Y, Then Coloplast Test product Z (Experimental): The subjects first test test product Y and after cross-over test product Z
  Interventions: Device: Coloplast Test product Y; Device: Coloplast Test product Z

INTERVENTIONS:
Device: Coloplast Test product Y — Coloplast Test product Y is a newly developed 2-piece convex ostomy appliance
  Other Names: Coloplast 2-piece Convex appliance Test product Y
Device: Coloplast Test product Z — Coloplast Test product Z is a newly developed 2-piece convex ostomy appliance
  Other Names: Coloplast 2-piece convex appliance test product Z

SUMMARY:
The aim of the current investigation is to develop new soft and more flexible 2-piece convex ostomy appliances

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and signed letter of authority.
2. Are at least 18 years of age and have full legal capacity.
3. Have had their ileostomy for at least 3 months.
4. Have used a 2-piece convex ostomy product during the last month.
5. Are willing and able to comply with investigation procedures.
6. Have an ileostomy with a diameter of 30 mm or less.
7. Have experienced leakage (seeping) under the baseplate at least 2 times during the last two weeks.

Exclusion Criteria:

1. Currently suffering from peristomal skin problems (i.e. bleeding or broken skin).
2. Currently receiving or have within the past 2 month received radio- and/or chemotherapy.
3. Currently receiving or have within the past month received local (peristomal area) or systemic steroid treatment.
4. Are pregnant or breastfeeding.
5. Have a loop ostomy (also called double-barrel or ostomy with two outlets).
6. Known hypersensitivity toward any of the test products.
7. Participating in other interventional clinical investigations or have previously participated in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Coloplast A/S
Locations (1):
- Coloplast A/S, Humlebæk, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited through the danish Coloplast database.
Period: Test Period 1
Arm/Group | First Coloplast Test Product Z; Then Coloplast Test Product Y | First Coloplast Test Product Y, Then Coloplast Test Product Z
Started | 10 | 10
Completed | 8 | 9
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Other | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Period: Test Period 2
Arm/Group | First Coloplast Test Product Z; Then Coloplast Test Product Y | First Coloplast Test Product Y, Then Coloplast Test Product Z
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Degree of Leakage
Description: The degree of leakage is measured using a 32-point scale developed by Coloplast A/S, where 0 represents No leakage (best possible outcome) and 32 points represents full-plate leakage (worst possible outcome).
  The degree of leakage was measured at each baseplate change.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: baseplate
Groups:
- Test Y; Test Z: Results from the subjects testing Coloplast Test Y
Arm/Group | Test Y | Test Z
Number analyzed (Participants) | 18 | 19
Number analyzed (baseplate) | 112 | 125
units on a scale | 5.0 (5.3) | 5.6 (5.7)

ADVERSE EVENTS:
Time Frame: The subjects were enrolled for 28+/- 3 days
Arm/Group | Test Y | Test Z
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 6/18 | 8/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Y (N=18) | Test Z (N=19)
Peristomal skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) — Related to device
Peristomal Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) — Related to device
Peristomal pain (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — related to device
broken peristomal skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Related to device
Pimple in peristomal area (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — related to device
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — not related to device
Fainted (General disorders) | 1 (1) | 0 (0) — not related to device
Headache (General disorders) | 1 (1) | 0 (0) — not related to device
Nausea (General disorders) | 1 (1) | 0 (0) — not related to device
wound on right arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — not related to device
Fungus infection in mouth (Infections and infestations) | 1 (1) | 0 (0) — not related to device
gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — not related to device
Vomit (Gastrointestinal disorders) | 0 (0) | 1 (1) — not related to device
chills in left side of bag and leg after applying the bag (General disorders) | 0 (0) | 1 (1) — 12 times
skin irritation on leg (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — where the bag cover the skin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes